CLINICAL TRIAL: NCT01045603
Title: A 3 Month Observational Prospective Patient Cohort Study of the Treatment of Breakthrough Pain in Cancer Patients With Instanyl®
Brief Title: Instanyl® Non-Interventional Study
Acronym: INIS
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: FT-1301-034-SP; U1111-1136-4251 (Registry Identifier: WHO)
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Breakthrough Cancer Pain
Keywords: Instanyl; non-interventional; breakthrough cancer pain; BTP; BTCP; Intranasal fentanyl spray

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to describe the use of Instanyl® (Intranasal fentanyl spray) in the treatment of breakthrough pain (BTP) in cancer patients by success of dose titration and distribution of dose strength. Data will be collected at three different time points over a 3 month period.

ELIGIBILITY:
* Adult cancer patients suffering from BTP
* Instanyl should be prescribed in accordance with the Summary of Product Characteristics (SPC) and none of the stated contradictions applies
* The decision to prescribe should be made independently of the study
* All patients must provide signed Informed Consent prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cancer patients (in- or out-patients) that are suffering from BTP who have not been treated with Instanyl for one month prior to Baseline.
Sampling Method: Non-Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2009-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Success of titration (Y/N), defined as reaching a maintenance dose | At week 4 and month 3 after baseline
Dose level of Instanyl® after titration, defined as the maintenance dose | At week 4 and month 3 after baseline

SECONDARY OUTCOMES:
Adverse Drug Reactions (ADR) | At week 4 and month 3 after baseline
Reason and time for Instanyl® termination | At week 4 and month 3 after baseline
Change in Instanyl® maintenance dose | At week 4 and month 3 after baseline
Change in level of background medication (standardised daily dose) | At week 4 and month 3 after baseline
Pain, pain relief and impact of pain of daily life | At baseline and week 4
Treatment satisfaction | At baseline and week 4

CONTACTS AND LOCATIONS:
Overall Officials: Nycomed Clinical Trial Operations, Study Chair — Headquarters
Locations (58):
- Denmark (4):
  - Investigational site, Copenhagen
  - Investigational site, Herning
  - Investigational site, Hillerød
  - Investigational site, Randers
- France (29):
  - Investigational site, Aix-en-Provence
  - Investigational site, Amiens
  - Investigational site, Argenteuil
  - Investigational site, Auxerre
  - Investigational site, Besançon
  - Investigational site, Blois
  - Investigational site, Bobigny
  - Investigational site, Bordeaux
  - Investigational site, Brest
  - Investigational site, Colmar
  - Investigational site, Eaubonne
  - Investigational site, Frelinghien
  - Investigational site, Grenoble
  - Investigational site, Lisieux
  - Investigational site, Lorient
  - Investigational site, Lyon
  - Investigational site, Montbéliard
  - Investigational site, Mulhouse
  - Investigational site, Nancy
  - Investigational site, Nantes
  - Investigational site, Orléans
  - Investigational site, Paris
  - Investigational site, Pierre-Bénite
  - Investigational site, Pontoise
  - Investigational site, Saint-Herblain
  - Investigational site, Strasbourg
  - Investigational site, Tarbes
  - Investigational site, Toulouse
  - Investigational site, Vandœuvre-lès-Nancy
- Investigational site, Athens, Greece
- Ireland (2):
  - Investigational site, Cork
  - Investigational site, Kilkenny
- Norway (9):
  - Investigational site, Bergen
  - Investigational site, Bodø
  - Investigational site, Fredrikstad
  - Investigational site, Haugesund
  - Investigational site, Kristiansand
  - Investigational site, Lørenskog
  - Investigational site, Oslo
  - Investigational site, Stavanger
  - Investigational site, Tromsø
- Sweden (6):
  - Investigational site, Alingsås
  - Investigational site, Stockholm
  - Investigational site, Sundsvall
  - Investigational site, Täby
  - Investigational site, Uppsala
  - Investigational site, Västervik
- United Kingdom (7):
  - Investigational site, Belfast
  - Investigational site, Lanarkshire
  - Investigational site, Luton
  - Investigational site, Manchester
  - Investigational site, Middlesex
  - Investigational site, Suffolk
  - Investigational site, Wiltshire